CLINICAL TRIAL: NCT06175065
Title: A Phase 2a Randomized, Doubled-Blind, Placebo-Controlled Trial to Evaluate Safety, Pharmacokinetics and Pharmacokinetic-Pharmacodynamic Relationships of RLS-0071 in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Safety, PK and PD Relationships of RLS-0071 in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLS-0071-204
Record Dates: First submitted 2023-11-29; First posted 2023-12-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
MeSH Terms: interventions — RLS-0071

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RLS-0071 (Experimental): Doses of RLS-0071, will be administered Q8H, three times a day, for at least 3 days and up to 5 days
  Interventions: Drug: RLS-0071
- Placebo (Placebo Comparator): Doses of Placebo for RLS-0071, will be administered Q8H, three times a day, for at least 3 days and up to 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLS-0071 — RLS-0071, will be administered as an IV infusion 10 mg/kg. Planned infusion duration is 8 minutes.
  Arms: RLS-0071
Drug: Placebo — Placebo control (commercial sterile saline), will be administered as an IV infusion. Planned infusion duration is 8 minutes.
  Arms: Placebo

SUMMARY:
AECOPD is a major cause of hospital admission and mortality. They contribute to long-term decline in lung function, physical capacity, and quality of life (QoL). RLS-0071 is a novel peptide being developed for the treatment of AECOPD. This study is designed to evaluate the safety and tolerability of RLS-0071 in the treatment of adults with moderate exacerbations of COPD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled trial in hospitalized participants with Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD) to evaluate the safety, tolerability, preliminary efficacy, PK, and PD of RLS-0071 compared to Placebo in the treatment of AECOPD. The dosing regimen will be 3 times a day for at least 3 days and up to 5 days total if still hospitalized. Participants will be followed for efficacy and safety for 30 and 60 days after the final dose. RLS-0071 or Placebo will be given as add-on therapy to SOC management for acute exacerbations of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized participants with a prior diagnosis of COPD including spirometry within the prior year documenting a postbronchodilator FEV1/FVC ≤ 0.7 and an FEV1

  ≤ 80%, and a clinician identified admitting diagnosis of AECOPD: acute increase in dyspnea, sputum volume or purulence - without other attributable cause.
* Participants must have a moderate exacerbation of COPD according to the Rome guidelines
* ≥ 10 pack-years smoking history.

Exclusion Criteria:

* Endotracheal intubation or mechanical ventilation.
* Participants with severe exacerbation of COPD according to the Rome guidelines
* Participants with signs and symptoms consistent with an alternative diagnosis for worsening of pulmonary status
* Interstitial lung disease.
* Current or prior history of asthma.
* Known hypersensitivity, allergy, or reaction to polyethylene glycol (PEG)
* Preexisting autoimmune disease: History of autoimmune disease and/or use of chronic steroids of >10mg/d (prednisone or equivalent) for more than 14 days prior to enrollment
* Current renal dialysis or renal dialysis planned or anticipated in the next 7 days.
* Has confounding medical conditions, including:

  1. diabetic coma,
  2. uncontrolled New York Heart Association Class IV congestive heart failure,
  3. uncontrolled angina,
  4. stroke or transient ischemic attack (TIA) within 4 weeks before study entry,
  5. clinically significant arrhythmias not controlled by medication, or
  6. idiopathic pulmonary fibrosis,
* Has a weight >120 kg at Screening.
* Known pregnancy, a positive pregnancy test at screening, or lactation for WOCBP.
* Has systemic immunosuppression/immune deficiency

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Day 1 to Day 60

SECONDARY OUTCOMES:
Time to reach maximum observed serum concentration (Tmax) for RLS-0071 | Day 1 and Day 3
Maximum Observed Serum Concentration (Cmax) for RLS-0071 | Day 1 and Day 3
Area Under the Curve From Time 0 to Infinity (AUC [0 - infinity]) for RLS-0071 | Day 1 and Day 3
Terminal Phase Elimination Half-Life (t1/2) for RLS-0071 | Day 1 and Day 3
Evaluate the change in plasma neutrophil counts from Day 0 up to Day 5. | Day 0 up to Day 5.
Evaluate the change from baseline in eosinophil counts from Day 0 up to Day 5. | Day 0 up to Day 5.
Evaluate the change from baseline in erythrocyte sedimentation rate from Day 0 up to Day 5. | Day 0 up to Day 5.
Evaluate the change in baseline in c-reactive protein in blood from Day 0 up to Day 5. | Day 0 up to Day 5.
Number of days participant was hospitalized (length of stay). | Day 1 - Day 60
Number of participants rehospitalized for COPD up to Day 60 | Day 1 to Day 60
Number of participants that progressed to mechanical ventilation | Day 1 - Day 5
Mortality rate of participants at 60 days after discharge | Day 1 to Day 60
Measure heart rate via beats per minute daily | Day 1 - Up to Day 5
Measure respiratory rate by measuring breaths per minute daily | Day 1 - Up to Day 5
Measure the % O2 saturation via pulse oximetry daily | Day 1 - Up to Day 5

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Site 02, St. Petersburg, Florida
  - Site 03, Glen Burnie, Maryland
  - Site 04, Omaha, Nebraska
  - Site 01, Philadelphia, Pennsylvania